CLINICAL TRIAL: NCT04075188
Title: Polypoidal Choroidal Vasculopathy in Pachychoroid: Aflibercept + PDT Combined Therapy
Brief Title: Treatment of Polypoidal Choroidal Vasculopathy in Pachychoroid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Principal Investigator, Salvatore Cillino, Head of the Ophthalmology Section of the Department of Biomedicine, Neurosciences and Advanced Diagnostic, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDT Aflibercept
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Choroidal Neovascularization; Choroid Disease
Keywords: pachychoroid; polypoidal choroidal vasculopathy; Aflibercept; photodynamic therapy; Swept source OCT
MeSH Terms: conditions — Choroidal Neovascularization; Choroid Diseases; Polypoidal Choroidal Vasculopathy | interventions — aflibercept; Verteporfin; Injections

STUDY DESIGN:
Intervention Model Description: Selected patients with both diagnosis of polypoidal choroidal vasculoparthy and pachychoroid will be treated with combined therapy consisting in photodynamic therapy and 3 intravitreal therapy of Aflibercept monthly
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined therapy (Experimental): Treatment consisting in photodynamic therapy (Verteporfin, 6 mg/m2 × Body Surface Area (BSA) = Total Drug Dose; Total Drug Dose ÷ 2.0 mg/mL = Volume of Reconstituted Verteporfin; 30 mL - Volume of Reconstituted Verteporfin = Volume of 5% dextrose in water. Light dose is 50 J/cm2 administered at an intensity of 600 mW/cm2. This dose is administered over 83 seconds) and 3 intravitreal therapy of Aflibercept (2 mg/0,05 ml)monthly, the first of which performed within 7 days from photodynamic therapy.
  Interventions: Drug: Aflibercept Injection

INTERVENTIONS:
Drug: Aflibercept Injection — Patients will be treated with combined therapy to determine the synergy of this treatment, causing anti- Vascular Endothelial Growth Factor (anti-VEGF) to block neovascular exudation and photodynamic therapy to close aneurismal vessel and reduce choroidal vascular congestion.
  Other Names: verteporfin for injection

SUMMARY:
This study will evaluate patients with diagnosis of polypoidal choroidal vasculopathy (PCV) in pachychoroid treated with combined therapy, consisting in photodynamic therapy (PDT) and 3 intravitreal therapy (IVT) of Aflibercept monthly. This is a single center, prospective case-series study. The investigators are going to evaluate Corrected Distance Visual Acuity (CDVA), disease activity, retinal and choroidal thicknesses and number of injection per year, during a twelve month follow up. The aim of this study is to verify if the combined therapy can act on the insult induced by the pachychoroid and on the neovascular lesion itself in this sub-population of patients with PCV in pachychoroid,

DETAILED DESCRIPTION:
This study evaluates patients with diagnosis of polypoidal choroidal vasculopathy (PCV) in pachychoroid treated with combined therapy, consisting in photodynamic therapy (PDT) and 3 intravitreal therapy (IVT) of Aflibercept monthly. Inclusion criteria are the presence of haemorrhagic or exudative PCV diagnosed by Optical Coherence Tomography (OCT) and Indocyanine Green Angiography (ICGA) and the mean central choroidal thickness > 250 µm. Exclusion criteria comprehend ocular comorbidity, previous cardiovascular events and different ocular surgical procedures form cataract surgery. Participants undergo a thorough ophthalmic assessment that included best corrected visual acuity (CDVA), slit lamp biomicroscopy and dilated funduscopic examination. OCT, OCT-Angiography (OCT-A), ICGA and Fluoresceine Angiography (FA) were performed for all patients. The 12-month follow-up foresee monthly revaluations of the above measurements, excluding FA, repeated only on clinical judgement. CDVA will be measured using LogMAR. Choroidal and retinal thicknesses will be automatically measured by digital software OCT- integrated (IMAGEnet). All patients will be treated with a loading dose of Aflibercept combined with PDT within the first 7 days of the first intravitreal therapy. The spot size is calculated by adding 1000 μm to the greater linear dimension of the lesion. No additional therapy will be performed during follow-up unless signs of reactivation.

ELIGIBILITY:
Inclusion Criteria:

* presence of haemorrhagic or exudative PCV diagnosed by OCT and ICGA
* Mean central choroidal thickness > 250 µm

Exclusion Criteria:

* ocular comorbidity
* previous cardiovascular events
* different ocular surgical procedures form cataract surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-07-13 (Actual)

PRIMARY OUTCOMES:
Corrected Distance Visual Acuity | twelve months
  measured in logMAR notation using Early Treatment of Diabetic Retinopathy Study charts (CC-100XP LCD System for ETDRS Chart display)
Disease Activity | twelve months
  measured as percentage of patients with subretinal or intraretinal fluid
Retinal Thickness | twelve months
  Central retinal thickness (1 mm central foveal thickness) and mean macular thickness (second and the third 6-mm grid including parafoveal and perifoveal macular area)
Choroidal thickness | twelve months
  Central choroidal thickness (1 mm central subfoveal thickness) and mean choroideal thickness (second and the third 6-mm grid including parafoveal and perifoveal choroidal area)

SECONDARY OUTCOMES:
Number of injections per year | twelve months
  Number of intravitreal injection administered in a year

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Cillino, MD PhD, Principal Investigator — AOUP Paolo Giaccone, Palermo
Locations (1):
- Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuzawa M, Mori R, Kawamura A. The origins of polypoidal choroidal vasculopathy. Br J Ophthalmol. 2005 May;89(5):602-7. doi: 10.1136/bjo.2004.049296. PMID 15834093
- [Background] Koh A, Lai TYY, Takahashi K, Wong TY, Chen LJ, Ruamviboonsuk P, Tan CS, Feller C, Margaron P, Lim TH, Lee WK; EVEREST II study group. Efficacy and Safety of Ranibizumab With or Without Verteporfin Photodynamic Therapy for Polypoidal Choroidal Vasculopathy: A Randomized Clinical Trial. JAMA Ophthalmol. 2017 Nov 1;135(11):1206-1213. doi: 10.1001/jamaophthalmol.2017.4030. PMID 28983556
- [Background] Wong TY, Ogura Y, Lee WK, Iida T, Chen SJ, Mitchell P, Gemmy Cheung CM, Zhang Z, Leal S, Ishibashi T; PLANET Investigators. Efficacy and Safety of Intravitreal Aflibercept for Polypoidal Choroidal Vasculopathy: Two-Year Results of the Aflibercept in Polypoidal Choroidal Vasculopathy Study. Am J Ophthalmol. 2019 Aug;204:80-89. doi: 10.1016/j.ajo.2019.02.027. Epub 2019 Mar 6. PMID 30849345
- [Background] Pang CE, Freund KB. Pachychoroid neovasculopathy. Retina. 2015 Jan;35(1):1-9. doi: 10.1097/IAE.0000000000000331. PMID 25158945
- [Background] Balaratnasingam C, Lee WK, Koizumi H, Dansingani K, Inoue M, Freund KB. Polypoidal Choroidal Vasculopathy: A Distinct Disease or Manifestation of Many? Retina. 2016 Jan;36(1):1-8. doi: 10.1097/IAE.0000000000000774. No abstract available. PMID 26414957
- [Background] Yanagi Y, Ting DSW, Ng WY, Lee SY, Mathur R, Chan CM, Yeo I, Wong TY, Cheung GCM. CHOROIDAL VASCULAR HYPERPERMEABILITY AS A PREDICTOR OF TREATMENT RESPONSE FOR POLYPOIDAL CHOROIDAL VASCULOPATHY. Retina. 2018 Aug;38(8):1509-1517. doi: 10.1097/IAE.0000000000001758. PMID 28704255